CLINICAL TRIAL: NCT00832312
Title: Intraarticular Ozone Therapy for Pain Control in Osteoarthritis of the Knee
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Because of technical problems (researcher moved to different city).
Sponsor: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Howard Tandeter, POB 653 Beer Sheva, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20080780
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Knee; Pain management; Ozone therapy; Intraarticular injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Agnosia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ozone-oxygen mixture (Experimental): 10 cc of an ozone-oxygen mixture with ozone concentration 10000 mcg/L (10 mcg/ml) injected into the knee joint
  Interventions: Other: ozone-oxygen mixture
- Saline (Placebo Comparator): Injection of 1cc of saline into the knee joint
  Interventions: Other: placebo (saline)

INTERVENTIONS:
Other: ozone-oxygen mixture — 10 cc of an ozone-oxygen mixture with ozone concentration 10000 mcg/L (10 mcg/ml)
  Arms: ozone-oxygen mixture
Other: placebo (saline) — Injection of 1cc of saline into the knee joint
  Arms: Saline

SUMMARY:
The purpose of this study is to determine whether an intraarticular injection of Ozone into the knee joint is an effective therapy for pain control in patients with osteoarthritis of the knee.

DETAILED DESCRIPTION:
Ozone, as a gas made of three atoms of oxygen with a cyclic structure, has been used as a medical therapy from the mid ninetieth century. Today, this therapy is a recognized modality in many European and Latin American nations for orthopedic problems, infections, ischemic diseases, and skin problems. However, despite of this wide use internationally, there is minimal mention of this treatment modality in the Anglo-American literature.

The present is the first of a series of studies planned to scientifically test the effectiveness of ozone as a main-stream therapy, introducing it to the Anglo-American literature. In this first study we will check whether intraarticular injections of Ozone into the knee joint are effective as a therapy for pain control in patients with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

- Osteoarthritis of knee

Exclusion Criteria:

* Positive rheumatologic serologic tests
* Cognitive impairment
* Adjacent osteomyelitis
* Bacteremia
* Hemarthrosis
* Impending (scheduled within days) joint replacement surgery
* Infectious arthritis
* Joint prosthesis
* Osteochondral fracture
* Periarticular cellulitis
* Poorly controlled diabetes mellitus
* Uncontrolled bleeding disorder or coagulopathy.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-08; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Pain control | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Howard B Tandeter, MD, Principal Investigator — Ben GurionUniversity
Locations (1):
- Ben Gurion University, Beersheba, Israel